CLINICAL TRIAL: NCT07143110
Title: LUNG-ROLL: Treatment Patterns and Cost of Illness of Lung Cancer in Canada
Acronym: LUNG-ROLL
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00044
Record Dates: First submitted 2025-05-30; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Lung Neoplasms
Keywords: Lung Neoplasms; Non-Small-Cell Lung; Small Cell Lung; Epidemiology; Treatment Patterns; Real-World
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Small Cell Lung Cancer (NSCLC)
- Small Cell Lung Cancer (SCLC)

SUMMARY:
LUNG-ROLL is a retrospective cohort study that will describe the contemporary treatment patterns, prevalence and incidence, patient demographic and clinical characteristics, clinical outcomes, and healthcare resource use/costs for patients with lung cancer in Canada (specifically, Alberta and Ontario) using administrative data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung cancer between January 1, 2018 and end of the Selection Period.
* Patient is 18 years of age or older on diagnosis date.
* Patient has at least 12 months of health insurance coverage prior to the diagnosis date.

Exclusion Criteria:

* Diagnosed with any other cancer in the 5-year period prior to January 1, 2018.
* Diagnosed with any other cancer concurrently (i.e., on the same date) as lung cancer diagnosis.
* Invalid or incomplete records for key variables (e.g., missing year of diagnosis, missing cancer type).
* Non-Ontario or non-Alberta resident on diagnosis date.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will comprise patients with lung cancer diagnosed after January 1, 2018 in the administrative databases for Alberta and Ontario.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment patterns | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Incidence and prevalence | Through study completion, an average of 1 year
Baseline demographic and clinical characteristics | Through study completion, an average of 1 year
Overall survival | Through study completion, an average of 6 months
Time to/on therapy | Through study completion, an average of 6 months
Attrition rates | Through study completion, an average of 1 year
Healthcare resource utilization (HCRU) | Through study completion, an average of 1 year
Direct healthcare costs | Through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: No